CLINICAL TRIAL: NCT06049628
Title: The Impact of FIFA 11+ Exercise Program on Isokinetic Muscle Strength and Balance on Adolescent Amateur Soccer Players.
Brief Title: The Impact of FIFA 11+ on Isokinetic Muscle Strength and Balance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: FIFA 11+
Record Dates: First submitted 2023-09-15; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-07

CONDITIONS: Injury Prevention
Keywords: adolescent; football; physical performance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FIFA 11+ group (Experimental): The experimental group will apply FIFA 11+ training 3 times a week for 9 weeks.
  Interventions: Behavioral: FIFA 11+ exercise program
- control group (Active Comparator): The control group members will be advised to continue their routine warm-up program 3 times a week for 9 weeks.
  Interventions: Behavioral: routine program

INTERVENTIONS:
Behavioral: FIFA 11+ exercise program — FIFA 11+ program; It consists of simple, easily remembered, and time-consuming, sport-specific exercises underlying fair play. The F 11+ consisted of 3 parts: the first part consisted of running exercises (part 1); the second part included six exercises, which were made up of three levels of difficulty and aimed at enhancing balance, strength, muscle control, and core stability (part 2). The final and the third part covered advanced running exercises (part 3) .
  Arms: FIFA 11+ group
Behavioral: routine program — This program consists of jogging, and stretching exercises.
  Arms: control group

SUMMARY:
FIFA 11+ program; It consists of simple, easily remembered, and time-consuming, sport-specific exercises underlying fair play. Although the FIFA 11+ program is a well-established warm-up protocol for injury prevention among football players, the performance improvement aspect of the program is not often discussed in the literature. The study's objective is to investigate the efficacy of the FIFA 11+ program on sports performance parameters such as dynamic balance, isokinetic muscle strength performance in adolescent amateur male football players.

DETAILED DESCRIPTION:
This study was planned in a randomized controlled experimental type. The footballers of a team from an amateur league will be included in the research. All participants will be tested at baseline and 9 weeks after baseline. The participants will be submitted to the following testing procedures: dynamic balance (Star Excursion Balance Test), muscle strength assessment (Isokinetic assessment). After the baseline measurements will be completed, the control group members will be advised to continue their regular warm-up program. This program consists of jogging and stretching exercises. The experimental group will complete the FIFA 11+ training, which consisted of six different types of running exercises; six exercises with three levels of increasing difficulty to improve the participants' strength, agility, core stability, eccentric control, etc.; and advanced running exercises, such as running across the pitch, bounding, planting, cutting. The FIFA 11+ will be applied to the experimental group 3 times a week for 9 weeks. The control group's warm-up duration will be matched to the experimental group's duration (20-25 min). This routine workout will perform 3 times a week for 9 weeks. At the end of 9 weeks, the evaluations will be repeated (Star Excursion Balance Test, Isokinetic assessment).

ELIGIBILITY:
Inclusion Criteria:

* ) To accept being a case study member
* ) Being in the 15-18 age range
* ) To be a soccer player in amateur league clubs with experience for at least one year
* ) Having no systemic diseases
* ) Having the necessary mental and physical activity level to be able to take and complete the tests

Exclusion Criteria:

* ) Refusing to be a member of a case study
* ) Having visual impairment and perceptual disorder at a severe level
* ) Having pain that prevents testing
* ) Having diseases with neurological dysfunction
* ) Footballers who stop playing active football during the study period and disrupt the training program by not participating in 3 exercises in a row
* ) Having an injury in the research process
* ) Having an injury in the last six months before the research

Ages: 15 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-12-30 (Actual)

PRIMARY OUTCOMES:
Isokinetic assessment | Baseline
  When assessing the football players in terms of strengths, frequently use isokinetic systems . Computer aided muscle-testing dynamometers are utilized for measuring muscle force and this provides us with an assessment of muscles and group of muscle in an isokinetic manner. Isokinetic muscle testing is conducted with a stable speed of angular motion yet variable resistance.
Isokinetic assessment | After the 9-week intervention
  When assessing the football players in terms of strengths, frequently use isokinetic systems . Computer aided muscle-testing dynamometers are utilized for measuring muscle force and this provides us with an assessment of muscles and group of muscle in an isokinetic manner. Isokinetic muscle testing is conducted with a stable speed of angular motion yet variable resistance
balance assessment | Baseline
  Dynamic postural control will be measured with the Star Excursion Balance Test (SEBT), which will be applied with a system of 8 lines. The foot will be placed in the center of the testing system to be bisected equally in the medial-lateral anteroposterior planes. SEBT is made up of 8 directions: anterior, anterolateral, lateral, posterolateral, posterior, posteromedial, medial, and anteromedial.
balance assessment | After the 9-week intervention
  Dynamic postural control will be measured with the Star Excursion Balance Test (SEBT), which will be applied with a system of 8 lines. The foot will be placed in the center of the testing system to be bisected equally in the medial-lateral anteroposterior planes. SEBT is made up of 8 directions: anterior, anterolateral, lateral, posterolateral, posterior, posteromedial, medial, and anteromedial.

CONTACTS AND LOCATIONS:
Overall Officials: büşra aydın erkılıç, MSc, Principal Investigator — Yeditepe University
Locations (1):
- Yeditepe University, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Ayala F, Pomares-Noguera C, Robles-Palazon FJ, Del Pilar Garcia-Vaquero M, Ruiz-Perez I, Hernandez-Sanchez S, De Ste Croix M. Training Effects of the FIFA 11+ and Harmoknee on Several Neuromuscular Parameters of Physical Performance Measures. Int J Sports Med. 2017 Apr;38(4):278-289. doi: 10.1055/s-0042-121260. Epub 2017 Feb 13. PMID 28192831